CLINICAL TRIAL: NCT06052098
Title: Transbronchial Versus Transthoracic Ablation for Early Stage Peripheral Lung Cancer: a Prospective, Randomized Controlled Trial
Brief Title: Transbronchial vs Transthoracic Ablation for Early-stage Peripheral Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Broncus Medical Co., Ltd. (Industry)
Collaborators: Shanghai Chest Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-I-RF-01
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-09

CONDITIONS: Stage IA Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transbronchial group (Experimental): Subjects receive bronchoscopy-guided RFA and undergo follow-up.
  Interventions: Device: The disposable pulmonary radiofrequency ablation catheter and pulmonary radiofrequency ablation system
- Transthoracic group (Experimental): Subjects receive CT-guided RFA and undergo follow-up.
  Interventions: Device: The disposable percutaneous radiofrequency ablation needle and pulmonary radiofrequency ablation system

INTERVENTIONS:
Device: The disposable pulmonary radiofrequency ablation catheter and pulmonary radiofrequency ablation system — Procedure: In combination with guided bronchoscopy and CBCT, the ablation catheter is placed in the target lesion. CBCT confirms the tool in the lesion, adjusts the position of the ablation catheter, and monitors the extent of ablation.
  Arms: Transbronchial group
Device: The disposable percutaneous radiofrequency ablation needle and pulmonary radiofrequency ablation system — Procedure: The ablation needle is punctured into the lesion under CT guidance. The extent of the ablation is monitored by CT.
  Arms: Transthoracic group

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of RFA through a transthoracic or transbronchial approach in the treatment of early-stage peripheral lung cancer.

DETAILED DESCRIPTION:
This study is designed as a prospective, randomized controlled trial with 110 participants, randomized in a 1:1 ratio to CT-guided RFA and bronchoscopy-guided RFA groups. The primary study endpoint is the complete ablation rate at 6 months post-ablation. Secondary study endpoints are technical success rate, complete ablation rate at 12 months post-ablation, local control rate at 1, 2, and 3 years post-ablation, progression free survival, overall survival, and safety. Demographic data, clinical baseline characteristics, CT follow-up data, and safety data will be collected and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years.
2. Primary peripheral lung cancer diagnosed by pathology, and preoperative staging reveals clinical stage T1N0M0, stage IA.
3. The planned ablation lesions are assessed to be amenable to CT-guided and bronchoscopy-guided ablation.
4. Assessed as inoperable or refused surgery, agree to undergo initial ablation therapy, and sign informed consent.

Exclusion Criteria:

1. Patients with platelet < 50 × 10 9/L, severe bleeding tendency and coagulation dysfunction that cannot be corrected in a short period of time.
2. Patients with severe pulmonary fibrosis and pulmonary hypertension.
3. Perilesional infection and radiation inflammation, puncture site skin infection is not well controlled, systemic infection, high fever > 38.5℃.
4. Patients with severe liver, kidney, heart, lung and brain dysfunction, severe anemia, dehydration and severe nutritional metabolism disorders that cannot be corrected or improved in a short period of time.
5. Patients with poorly controlled malignant pleural effusion.
6. Anticoagulation therapy and/or antiplatelet agents (except novel oral anticoagulants such as dabigatran and rivaroxaban) are discontinued for less than 5~7 days before ablation.
7. Eastern Cooperative Oncology Group (ECOG) score > 2.
8. Combined with other tumors with extensive metastasis, expected survival < 6 months.
9. Patients with episodic psychosis.
10. Patients with implantable electronic devices (such as pacemaker or defibrillator).
11. Pregnant women, or patients who have pregnancy plans during the study.
12. Participation or ongoing participation in another clinical study within the past 30 days.
13. Other situations that the investigator deems inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Complete ablation rate at 6 months after ablation | 6 months
  It is defined as the proportion of lesions with complete ablation to all ablated lesions at 6 months after ablation.

SECONDARY OUTCOMES:
Technical success rate | Immediately after ablation
  It is defined as the proportion of lesions which the ablation needle reached and successfully ablated to all lesions intended for ablation.
Complete ablation rate 12 months after ablation | 12 months
  It is defined as the proportion of lesions with complete ablation to all ablated lesions at 12 months after ablation.
Local control rate at 1 year, 2 years and 3 years after ablation | 1 year, 2 years and 3years
  It is defined as the proportion of lesions with complete ablation and incomplete ablation to all ablated lesions at 1 year, 2 years, and 3 years after ablation.
Progression free survival (PFS) | 3 years
  It is defined as the duration from the ablation to the first occurrence of disease progression or the death of the subject.
Overall survival (OS) | 3 years
  It is defined as the total time from the ablation to the death of the subject.
Safety | 12 months
  To assess the incidence of device- or procedure-related (serious) adverse events occurring during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No